CLINICAL TRIAL: NCT00000220
Title: Gradual Vs. Rapid Buprenorphine Detoxification
Brief Title: Gradual Vs. Rapid Buprenorphine Detoxification - 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06969-2; R01-06969-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-09

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine an optimal detoxification dose reduction schedule with buprenorphine.

ELIGIBILITY:
Please contact site for information.

Ages: 33 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1991-06; Study Completion 2001-07

PRIMARY OUTCOMES:
Drug use
Retention
Observed withdrawal rating
Opioid agonist rating
Opioid antagonist rating

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] Amass L, Bickel WK, Higgins ST, Hughes JR. A preliminary investigation of outcome following gradual or rapid buprenorphine detoxification. J Addict Dis. 1994;13(3):33-45. doi: 10.1300/j069v13n03_04. PMID 7734458